CLINICAL TRIAL: NCT05422352
Title: Role of Carnosine in Combination With Vitamin B Complex in Preventing the Progression of Diabetic Neuropathy in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahitab Hany Ahmed, Principle investigator (Assistant lecturer of clinical pharmacy department ), Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Carnosine Diabetic neuropathy
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Neuropathies
Keywords: Carnosine; diabetic neuropathy; oxidative stress; inflammation; Nerve conduction; type 2 diabetes; hyperglycemia; neopterin; nerve growth factor
MeSH Terms: conditions — Diabetic Neuropathies; Inflammation; Diabetes Mellitus, Type 2; Hyperglycemia; Hereditary Sensory and Autonomic Neuropathies | interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: intervention study clinical trial
Masking Description: intervention clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention Group (Experimental): Patients who will receive carnosine supplementation + Vitamin B complex two tablets per day
  Interventions: Dietary Supplement: Carnosine
- Control group (No Intervention): Patients will receive only Vitamin B Complex two tablets per day

INTERVENTIONS:
Dietary Supplement: Carnosine — Patients who will receive carnosine supplementation 500mg capsules (Now foods) in combination with Vitamin B complex (B1+B6+B12, 150 mg+100 mg+1 mg, respectively, Neurovit, European Egyptian Pharm. Ind., Egypt), two tablets per day
  Arms: intervention Group

SUMMARY:
Evaluation of the influence of oral administration of carnosine in combination with vitamin B Complex in preventing the progression of diabetic neuropathy in type 2 diabetes patients.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) is considered the most common chronic complication of diabetes mellitus, with an incidence rate of about 50%.

DPN is a group of clinical syndromes that affects single or combined regions in the nervous system and is considered one of the microvascular complications that affect greatly the quality of life of patients due to pain and frequency of hospitalization.

DPN commonly develops silent without symptoms in the early stages and when symptoms start appearing only a few effective therapies are available and that is what causes significant patient suffering and societal burden.

Those mechanisms of pain and treatment remain challenging and are restricted by variable efficacy and side effects of therapies and intensification of glycemic control remain the cornerstone for the prevention or delay of DPN.

Lately, it has been proven that long-term low-grade inflammation has an important role in DPN pathogenesis. Clinical trials in DPN patients with pain and without pain showed that the DPN with pain group had higher inflammation markers.

In addition, DPN patients with pain had more increased cytokine levels compared with DPN patients without pain. Besides the correlation between abnormalities in nerve fibers and the rise in interleukin (IL)-6 and IL-10.

Moreover, Oxidative stress plays an important role in the development of diabetic neuropathy a reactive oxygen species (ROS) increases the progression of nerve fiber damage and dysfunction.

Those reactive oxygen species are capable of destroying the lipids found in the myelinated structures of nerves resulting in axon loss and disturbance in the microvasculature of the peripheral nervous system.

Antioxidants are available endogenously as a normal defense mechanism of the cell or obtained exogenously from diet and could play an important role in the progression of damage to the neurons in Diabetic neuropathy.

Carnosine, a naturally-occurring dipeptide (β-alanyl-L-histidine) first described in 1900 by Gulewitsch and Amiradzibi, is found predominantly in post-mitotic tissues (e.g. brain and innervated muscle) of vertebrates.

Carnosine is claimed to decrease oxygen-free-radical mediated damage to cellular macromolecules either by chelating divalent cations or scavenging hydroxy radicals with its imidazole moiety. Free-radical damage is not the only process to affects the structure of proteins and nucleic acids.

Furthermore, previous studies proved the neuroprotective action of carnosine with its anti-inflammatory and antioxidant properties.

Moreover, another study highlighted the use of carnosine as a supportive treatment against neurotoxins.

Also, Carnosine has been shown to protect cultured neurons from oxygen-glucose deprivation and to exhibit neuroprotective properties in animal models of global and cerebral ischemia

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes Patients as per ADA criteria.
* Patients were showing clinical signs of Diabetic neuropathy verified by a neurologist and confirmed by a score ≥7 on the MNSI questionnaire (Michigan Neuropathy Screening Instrument), with abnormal nerve conduction measurement.
* Patients on a regular visit to the clinic.

Exclusion Criteria:

* Patients with neuropathy of non-diabetic origin were excluded.
* Patients with a BMI of 40 kg/m2 or more and those pregnant or breastfeeding were also excluded

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Neopterin biomarker | 3 months
  Neopterin, a marker of inflammation and cellular immune response, is elevated in conditions of T-cell or macrophages activation. Diabetic peripheral neuropathy (DPN) is associated with inflammatory/immune processes therefore Investigators hypothesized that it will decrease after intervention
malondialdehyde biomarker | 3 months
  it is oxidative stress marker that increases in the lipid peroxidation and inflammation happening during diabetic neuropathy and investigators hypothesized that it will decrease after intervention
Nerve Growth Factor | 3 months
  a neurotrophic factor and neuropeptide primarily involved in the regulation of growth, maintenance, proliferation, and survival of certain target neurons and investigathypothesized its increase after intervention
Nerve Growth Factor | 3 months
  a neurotrophic factor and neuropeptide primarily involved in the regulation of growth, maintenance, proliferation, and survival of certain target neurons and investigators hypothesized its increase after intervention

CONTACTS AND LOCATIONS:
Overall Officials: H F Salem, Professor, Study Chair — Beni-Suef University
Locations (1):
- Beni Suef University faculty of pharmacy, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hipkiss AR. Glycation, ageing and carnosine: are carnivorous diets beneficial? Mech Ageing Dev. 2005 Oct;126(10):1034-9. doi: 10.1016/j.mad.2005.05.002. PMID 15955546
- [Result] Oyenihi AB, Ayeleso AO, Mukwevho E, Masola B. Antioxidant strategies in the management of diabetic neuropathy. Biomed Res Int. 2015;2015:515042. doi: 10.1155/2015/515042. Epub 2015 Mar 2. PMID 25821809
- [Result] Edwards JL, Vincent AM, Cheng HT, Feldman EL. Diabetic neuropathy: mechanisms to management. Pharmacol Ther. 2008 Oct;120(1):1-34. doi: 10.1016/j.pharmthera.2008.05.005. Epub 2008 Jun 13. PMID 18616962
- [Result] Tesfaye S, Selvarajah D. Advances in the epidemiology, pathogenesis and management of diabetic peripheral neuropathy. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:8-14. doi: 10.1002/dmrr.2239. PMID 22271716
- [Result] Vinik A I, "Diabetic Neuropathies," Contemp. Endocrinol. Controv. Treat. Diabetes Clin. Res. Asp.(2000), 109-134.
- [Result] Callaghan BC, Cheng HT, Stables CL, Smith AL, Feldman EL. Diabetic neuropathy: clinical manifestations and current treatments. Lancet Neurol. 2012 Jun;11(6):521-34. doi: 10.1016/S1474-4422(12)70065-0. Epub 2012 May 16. PMID 22608666
- [Result] Shakher J, Stevens MJ. Update on the management of diabetic polyneuropathies. Diabetes Metab Syndr Obes. 2011;4:289-305. doi: 10.2147/DMSO.S11324. Epub 2011 Jul 21. PMID 21887102
- [Result] Jin HY, Park TS. Role of inflammatory biomarkers in diabetic peripheral neuropathy. J Diabetes Investig. 2018 Sep;9(5):1016-1018. doi: 10.1111/jdi.12794. Epub 2018 Jan 22. PMID 29277966
- [Result] Doupis J, Lyons TE, Wu S, Gnardellis C, Dinh T, Veves A. Microvascular reactivity and inflammatory cytokines in painful and painless peripheral diabetic neuropathy. J Clin Endocrinol Metab. 2009 Jun;94(6):2157-63. doi: 10.1210/jc.2008-2385. Epub 2009 Mar 10. PMID 19276232
- [Result] Hipkiss AR, Michaelis J, Syrris P. Non-enzymatic glycosylation of the dipeptide L-carnosine, a potential anti-protein-cross-linking agent. FEBS Lett. 1995 Aug 28;371(1):81-5. doi: 10.1016/0014-5793(95)00849-5. PMID 7664889
- [Result] Tsai SJ, Kuo WW, Liu WH, Yin MC. Antioxidative and anti-inflammatory protection from carnosine in the striatum of MPTP-treated mice. J Agric Food Chem. 2010 Nov 10;58(21):11510-6. doi: 10.1021/jf103258p. Epub 2010 Oct 6. PMID 20925384